CLINICAL TRIAL: NCT05257213
Title: Intrauterine Adhesions Prevention: the Use of Heparin Solution Compared to Application of Anti-adhesion Barrier Gel After Operative Hysteroscopy
Brief Title: Heparin Solution Versus Anti-adhesion Barrier Gel for Intrauterine Adhesions Prevention After Operative Hysteroscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nadezhda Women's Health Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3/11022022
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Intrauterine Adhesion
Keywords: operative hysteroscopy; heparin; anti-adhesion barrier gel; intrauterine adhesion; hyaluronic acid
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Intervention Model Description: Comparison between two active intrauterine treatments administered immediately post surgery
Who Masked: Participant
Masking Description: Patients will be under general anaesthesia during surgical procedure when the allocated treatment will be administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Heparin solution (Active Comparator): Administration of 3 ml heparin solution into the uterine cavity via a syringe immediately post operative hysteroscopy.
  Interventions: Drug: Heparin solution
- Anti-adhesion barrier gel (Active Comparator): Intrauterine application of 2 ml biodegradable anti-adhesion barrier gel immediately post operative hysteroscopy.
  Interventions: Drug: Anti-adhesion barrier gel

INTERVENTIONS:
Drug: Heparin solution — 3 ml saline solution containing 5000 IU heparin.
  Other Names: HEP
  Arms: Heparin solution
Drug: Anti-adhesion barrier gel — 2 ml biodegradable barrier gel containing sodium hyaluronate (10 mg/ml), sodium chloride (8.5 mg/ml), disodium hydrogen phosphate (0.34mg/ml), sodium dihydrogen phosphate (0.14 mg/ml) and water for injection (QS to weight).
  Other Names: AAB
  Arms: Anti-adhesion barrier gel

SUMMARY:
The aim of this study is to compare the efficacy of intrauterine application of heparin solution to the use of hyaluronic acid barrier gel for the prevention of intrauterine adhesion formation after operative hysteroscopy.

DETAILED DESCRIPTION:
In this trial the investigators aim to evaluate and compare the effect of heparin solution to anti-adhesive hyaluronic barrier gel administration immediately after operative hysteroscopy on post-surgical complications (incidence, extent and severity of intrauterine adhesions, abnormal menstrual cycle pattern) and fertility.

Patients undergoing operative hysteroscopy will be identified and invited to participate in the trial. At 4 to 8 weeks after the initial surgery, a follow-up, diagnostic hysteroscopy will be performed to identify indications for subsequent operative procedure and classify intrauterine adhesions according to extent of uterine cavity affected and type of formation found. Data on subsequent persistent irregular menstrual bleeding and pregnancy success up to 12 months following treatment will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* female sex
* indication for operative hysteroscopy including one or more of the following:
* infertility,
* irregular bleeding,
* oligo-/amenorrhea,
* Asherman syndrome,
* G0-G3 fibroids,
* dysmorphic uterus.

Exclusion Criteria:

* ongoing pregnancy,
* genital cancer,
* pelvic inflammatory disease,
* excessive uterine bleeding.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2026-02-14 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of patients with post-operative intrauterine adhesion formation | 4 to 8 weeks post treatment
  Incidence and severity of intrauterine adhesions identified at follow-up diagnostic hysteroscopy as assessed according to Valle and Sciarra's classification of intrauterine synaechia
Number of patients with need for subsequent operative hysterectomy | 4 tot 8 weeks post treatment
  Pathological findings at second-look hysteroscopy taken as indication for successive uterine surgery
Number of patients with persistent irregular menstrual bleeding | up to 12 months post treatment
  Recurring abnormal menstrual cycle patterns identified post initial surgery

SECONDARY OUTCOMES:
Number of patients with fertility improvement | up to 12 months post treatment
  Successful pregnancy post surgical procedure

CONTACTS AND LOCATIONS:
Locations (2):
- Bulgaria (2):
  - Nadezhda Women's Health Hospital, Sofia, Sofia
  - Nadezhda Women's Health Hospital, Sofia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Healy MW, Schexnayder B, Connell MT, Terry N, DeCherney AH, Csokmay JM, Yauger BJ, Hill MJ. Intrauterine adhesion prevention after hysteroscopy: a systematic review and meta-analysis. Am J Obstet Gynecol. 2016 Sep;215(3):267-275.e7. doi: 10.1016/j.ajog.2016.05.001. Epub 2016 May 10. PMID 27173082
- [Background] Valle RF, Sciarra JJ. Intrauterine adhesions: hysteroscopic diagnosis, classification, treatment, and reproductive outcome. Am J Obstet Gynecol. 1988 Jun;158(6 Pt 1):1459-70. doi: 10.1016/0002-9378(88)90382-1. PMID 3381869
- [Background] Nappi C, Di Spiezio Sardo A, Greco E, Guida M, Bettocchi S, Bifulco G. Prevention of adhesions in gynaecological endoscopy. Hum Reprod Update. 2007 Jul-Aug;13(4):379-94. doi: 10.1093/humupd/dml061. Epub 2007 Apr 23. PMID 17452399
- [Background] van Wessel S, Hamerlynck T, Schutyser V, Tomassetti C, Wyns C, Nisolle M, Verguts J, Colman R, Weyers S, Bosteels J. Anti-adhesion Gel versus No gel following Operative Hysteroscopy prior to Subsequent fertility Treatment or timed InterCourse (AGNOHSTIC), a randomised controlled trial: protocol. Hum Reprod Open. 2021 Feb 16;2021(1):hoab001. doi: 10.1093/hropen/hoab001. eCollection 2021. PMID 33623830
- [Background] Lee WL, Liu CH, Cheng M, Chang WH, Liu WM, Wang PH. Focus on the Primary Prevention of Intrauterine Adhesions: Current Concept and Vision. Int J Mol Sci. 2021 May 13;22(10):5175. doi: 10.3390/ijms22105175. PMID 34068335